CLINICAL TRIAL: NCT01955915
Title: Characterization of Small Choroidal Tumors Using Functional Optical Coherence Tomography
Brief Title: Blood Vessel Patterns in Small Choroidal Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Alison Skalet, Alison Skalet, MD, PhD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: IRB00009475; IRB#00009475 (Other: OHSU Institutional Review Board)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Small Posterior Choroidal Tumors
Keywords: choroid; tumor; OCT; malignant melanoma
MeSH Terms: conditions — Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Choroidal Tumor Group: 15 patients diagnosed with small posterior choroidal tumors will be considered and evaluated for enrollment into this study

SUMMARY:
The purpose of this study is to see if mapping blood vessel patterns with optical coherence tomography (OCT) will help identify life-threatening choroidal tumors in their early stages and improve overall patient survival through early detection.

DETAILED DESCRIPTION:
Uveal melanomas are melanocytic tumors that arise in the pigmented tissues of the eye: the iris, ciliary body, and choroid. Iris melanomas rarely metastasize (spread to other tissues or organs). In contrast, uveal melanomas arising in the ciliary body and choroid are highly malignant (cancerous and invasive to other tissues or organs). Despite having excellent local tumor control rates, uveal melanoma remains a life-threatening cancer, and even eye-sparing therapy with radiation treatment often leads to significant loss of vision. Therefore patients diagnosed with uveal melanoma must cope with not only a life-threatening illness, but also the frightening prospect of significant vision loss. Choroidal melanomas located in the posterior pole, an anatomical area of the eye which includes the optic nerve and macula (central retina), are of particular concern with regards to visual outcome, as radiation treatment to these areas for even the smallest of tumors is often associated with severe vision loss. The accurate diagnosis and treatment of small choroidal melanomas is critical to patient survival. When tumors with metastatic potential are recognized and treated at an early stage, survival prognosis improves dramatically.

The purpose of this study is to learn if malignant (life-threatening) choroidal tumors versus benign (non-life-threatening) tumors will show distinct blood vessel patterns using functional optical coherence tomography (OCT) angiography. Angiography is the mapping of blood vessels. The investigators believe that OCT angiography can provide data which may help in identifying life-threatening tumors at the earliest stages and improve overall survival for patients with this type of melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than age 18 with small (< 3mm) choroidal tumors located within the posterior pole region which can be imaged using OCT technology. Subjects with benign-appearing and malignant-appearing lesions meeting these criteria will be enrolled.

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging.
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
* Women who are pregnant or lactating at the time of enrollment due to unknown safety of fluorescein angiography. Women that become pregnant during the course of the study may remain enrolled; however, flurorescein and ICG angiography will not be performed until they are no longer pregnant or nursing an infant.
* Patients receiving treatment for uveal melanomas will be excluded from the longitudinal natural history portion of this study, but may enroll for a single study visit prior to treatment of their melanoma. They will then be eligible to enroll in IRB 9501, which will follow radiation-treated patients longitudinally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will measure blood vessel pattern/flow changes in 15 patients with small posterior choroidal tumors.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Blood vessel patterns in small choroidal tumors | 24 months
  To determine if identifying early changes in blood vessel patterns will aid in early diagnosis and treatment of potentially aggressive choroidal tumors. This will be assessed using functional OCT angiography technology.

CONTACTS AND LOCATIONS:
Overall Officials: Alilson Skalet, MD, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided